CLINICAL TRIAL: NCT05346354
Title: A Phase 2/3, Open-label, Historical-controlled, Single-arm, Multicenter Study to Evaluate the Efficacy, Pharmacokinetics, Pharmacodynamics, and Safety of Ravulizumab in Children and Adolescents With Aquaporin-4 Antibody Positive (AQP4-Ab [+]) Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: Efficacy and Safety Study of Ravulizumab IV in Pediatric Participants With NMOSD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-NMO-317
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica Spectrum Disorder; Ravulizumab; ALXN1210; CNS Autoimmune Disorders; NMO; NMOSD
MeSH Terms: conditions — Neuromyelitis Optica | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ravulizumab (Experimental): During the Primary Treatment Period, all participants will receive weight-based dosing of ravulizumab IV for a total of 50 weeks of treatment.
  During the Extension Period, participants will continue to receive weight-based dosing of ravulizumab IV for up to 104 weeks.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Participants will receive a weight-based loading dose of ravulizumab on Day 1, followed by weight-based maintenance treatment with ravulizumab on Day 15 and every 8 weeks (q8w) after or once every 4 weeks (q4w) depending on weight.
  During the Extension Period, participants will continue to receive weight-based maintenance doses of ravulizumab IV on Day 351 and q8w or q4w, depending on weight.
  Other Names: ALXN1210; Ultomiris

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of ravulizumab in pediatric participants with Neuromyelitis Optica Spectrum Disorder (NMOSD).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be anti-AQP4 Ab-positive and have a diagnosis of NMOSD as defined by the 2015 international consensus diagnostic criteria.
* Complement inhibitor treatment-naïve participants must have had at least 1 attack or relapse in the last 12 months prior to the Screening Period.
* Expanded Disability Status Scale (EDSS) score ≤ 7.
* Eculizumab-experienced participants must be clinically stable per Investigator for 30 days and have been treated with eculizumab in Study ECU-NMO-303 for at least 90 days prior to screening with no missed doses within 2 months prior to Day 1.
* Participants who enter the study receiving supportive IST(s) (eg, corticosteroid, azathioprine [AZA], mycophenolate mofetil [MMF], methotrexate [MTX], tacrolimus [TAC], cyclosporin [CsA], or cyclophosphamide [CYC]) for the prevention of relapse, either in combination or monotherapy, must be on a stable dosing regimen of adequate duration prior to Screening and remain on a stable dosing regimen during the Screening Period.
* To reduce the risk of meningococcal infection (Neisseria meningitidis), all participants must be vaccinated against meningococcal infection.
* Documented vaccination for Hib and S pneumoniae at least 14 days prior to Day 1 according to national/local guidelines for the applicable age group.

Exclusion Criteria:

* Use of rituximab within 3 months prior to screening.
* Currently treated with a biologic medications (other than eculizumab) that may affect immune system functioning, or has stopped treatment with a biologic medication that may affect immune system functioning, and 5 half lives of the medication have not elapsed by the time of the Screening Visit.
* Use of intravenous immunoglobulin (IVIg) or plasma exchange (PE) within 3 weeks prior to Screening.
* Participation in another investigational drug or investigational device study (other than Study ECU-NMO-303) within 5 half lives of that investigational product (if known) or 30 days before initiation of the first dose of study drug, whichever is longer.
* Use of immunomodulatory therapies for multiple sclerosis within 3 months prior to Screening.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2029-04-02 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Annualized Relapse Rate at Week 50 | Baseline, Week 50
Time to First Adjudicated On-trial Relapse through Week 50 | Baseline through Week 50

SECONDARY OUTCOMES:
Change From Baseline in Expanded Disability Status Scale Score At Week 50 | Baseline, Week 50
  The score ranges are 0 to 10, higher score indicates worse outcome.
Change From Baseline in Hauser Ambulation Index at Week 50 | Baseline, Week 50
  The score ranges are 0 to 9, higher score indicates worse outcome.
Change From Baseline in Visual Acuity at Week 50 | Baseline, Week 50
Change From Baseline in Confrontational Visual Fields at Week 50 | Baseline, Week 50
Change From Baseline in Color Vision at Week 50 | Baseline, Week 50
Serum Ravulizumab Concentration | Predose and postdose (at end of infusion) on Day 1, Weeks 2, 10, 18, 26, and 42, and predose on Week 50
Change from Baseline in Free Serum Complement Component 5 (C5) Concentration Over Time Through Week 50 | Baseline through Week 50

CONTACTS AND LOCATIONS:
Locations (21):
- United States (6):
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Miami, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Durham, North Carolina
  - Research Site, Philadelphia, Pennsylvania
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (3):
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Marseille
  - Research Site, Montpellier
- Germany (2):
  - Research Site, Bochum
  - Research Site, Giessen
- Italy (4):
  - Research Site, Catania
  - Research Site, Chieti
  - Research Site, Gallarate
  - Research Site, Roma
- Research Site, Yokohama, Japan
- Research Site, Goyang-si, South Korea
- Research Site, Esplugues de Llobregat, Spain

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.